CLINICAL TRIAL: NCT00089609
Title: A Phase II Trial of Docetaxel, Thalidomide, Prednisone and Bevacizumab in Patients With Androgen-Independent Prostate Cancer
Brief Title: Docetaxel, Thalidomide, Prednisone, and Bevacizumab to Treat Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040257; 04-C-0257; NCT00091364 (obsolete NCT alias)
Record Dates: First submitted 2004-08-06; First posted 2004-08-09 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Prostatic Neoplasms
Keywords: Hormones; Angiogenesis; Markers; Tumor; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Docetaxel; Thalidomide; Prednisone; Bevacizumab; Amplified Fragment Length Polymorphism Analysis; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Main cohort - Prostate Cancer (Experimental): Docetaxel 75 mg/m^2 intravenously over 60 minutes on cycle 1 day 1 repeated every 21 days. Thalidomide 200 mg by mouth daily throughout the cycle. Prednisone 10 mg by mouth daily throughout the cycle. Bevacizumab 15 mg/kg intravenously on cycle 1 day 1 every 21 days.
  Interventions: Drug: Docetaxel; Drug: Thalidomide; Drug: Prednisone; Biological: bevacizumab; Genetic: polymorphism analysis; Other: immunoenzyme technique; Other: laboratory biomarker analysis; Other: pharmacological study
- Expansion cohort - Prostate Cancer (Experimental): Docetaxel 75 mg/m^2 intravenously over 60 minutes and Bevacizumab 15 mg/kg intravenously was given for 2 cycles. After two cycles Prednisone 10 mg by mouth daily and Thalidomide 200 mg by mouth daily was added.
  Interventions: Drug: Docetaxel; Drug: Thalidomide; Drug: Prednisone; Biological: bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m^2 intravenously over 60 minutes on cycle 1 day 1 repeated every 21 days.
  Other Names: Taxotere
Drug: Thalidomide — Thalidomide 200 mg by mouth daily throughout the cycle.
  Other Names: Thalomid
Drug: Prednisone — Prednisone 10 mg by mouth daily throughout the cycle.
  Other Names: Deltasone
Biological: bevacizumab — Bevacizumab 15 mg/kg intravenously on cycle 1 day 1 every 21 days.
  Other Names: Avastin
Genetic: polymorphism analysis — Two buffy coat tubes (two 7mL blue tiger top tubes) will be obtained and wrapped in foil when the patient enters onto the study. DNA (deoxyribonucleic acid) will be isolated only for the purpose of genotype analysis of enzymes with putative relevance for docetaxel or thalidomide disposition.
  Arms: Main cohort - Prostate Cancer
Other: immunoenzyme technique — The PBMC (peripheral blood mononuclear cells) of patients will be analyzed pre-treatment and post cycle 2 for any changes in the function of regulatory T cells. The following analysis will be performed: flow cytometry analysis, CD4 CD25 T cell enrichment, and immunosuppression assay.
  Arms: Main cohort - Prostate Cancer
Other: laboratory biomarker analysis — Serum and urine samples will be collected at baseline and monthly to measure VEGF (vascular endothelial growth factor) levels.
  Arms: Main cohort - Prostate Cancer
Other: pharmacological study — Plasma concentrations of docetaxel and thalidomide will be determined to assess interactions between docetaxel (and thalidomide) and the concomitant therapy.The analysis will be performed using a validated method based on liquid chromotography with mass-spectrometric detection.
  Arms: Main cohort - Prostate Cancer

SUMMARY:
This is a Phase II study of docetaxel, bevacizumab, prednisone and thalidomide in patients with androgen independent metastatic prostate cancer who are previously untreated with chemotherapy. The primary objective of this study is to determine if the combination of docetaxel, thalidomide and bevacizumab is able to be associated with a sufficiently high proportion of patients with a prostate-specific antigen (PSA) response to be worthy of further investigation in metastatic prostate cancer. We will also be looking at multiple secondary endpoints. These will include possible pharmacokinetic interactions among the study agents, potential correlation between patient genotype and efficacy of treatment. We will also be looking for circulating tumor cells in blood before and after treatment. Additionally we will be monitoring the tolerability of the regimen and survival duration as endpoints as well. We hope to use this trial to build on the promising results seen in our thalidomide/docetaxel protocol where there was a significant PSA decline and a trend toward survival benefit.

DETAILED DESCRIPTION:
This is a Phase II study of docetaxel, bevacizumab, prednisone and thalidomide in patients with androgen independent metastatic prostate cancer who are previously untreated with chemotherapy. The primary objective of this study is to determine if the combination of docetaxel, thalidomide and bevacizumab is able to be associated with a sufficiently high proportion of patients with a PSA response to be worthy of further investigation in metastatic prostate cancer. We will also be looking at multiple secondary endpoints. These will include possible pharmacokinetic interactions among the study agents, potential correlation between patient genotype and efficacy of treatment. We will also be looking for circulating endothelial cells in blood before and after treatment. Additionally we will be monitoring the tolerability of the regimen, time to disease progression, and survival duration as endpoints as well. We hope to use this trial to build on the promising results seen in our thalidomide/docetaxel protocol where there was a significant PSA decline and a trend toward survival benefit.

ELIGIBILITY:
* INCLUSION CRITERIA:

Androgen-independent metastatic adenocarcinoma of the prostate defined as progressive metastatic disease while on gonadotropin releasing hormone (GnRH) agonists or post surgical castration

Histopathological documentation of prostate cancer confirmed in the National Cancer Institute (NCI) Laboratory of Pathology at the National Institutes of Health, the Pathology Department at Walter Reed Medical Center or the Pathology Department at National Naval Medical Center, prior to starting this study. In addition, patients whose slides are lost or unavailable will be eligible for the study if they provide documentation of prostate cancer and if they meet criteria of clinically progressive prostate cancer as outlined in section 3.1.1.3.

Clinically progressive prostate cancer documented prior to entry. Progression must be documented by at least one of the following parameters:

* Two consecutively rising prostate-specific antigen (PSA) levels. The first rising PSA must be a minimum of one week from a reference value. It is recognized that PSA fluctuations are such that the confirmatory PSA value might be less than the previous one. In these cases, that patient would still be eligible provided the next PSA was greater than the first rising PSA value. Patients must have PSA greater than or equal to 5.0.
* At least one new lesion on bone scan.
* Progressive measurable disease.

Patients must have undergone bilateral surgical castration or must continue on GNRH agonist.

Those patients receiving an anti-androgen agent and are entering the trial due to a rise in PSA must demonstrate a continued rise in PSA 4 weeks after stopping flutamide and 6 weeks after stopping bicalutamide or nilutamide.

Patients may not have received any chemotherapy for metastatic prostate cancer

Age greater than or equal to 18 years

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Life expectancy of greater than 3 months

Patients must have adequate organ and marrow function as defined below:

Leukocytes- greater than or equal to 3,000/microliter

Absolute neutrophil count- greater than or equal to 1,500/microliter

Platelets- greater than or equal to 100,000/microliter

Hemoglobin- greater than or equal to 8.0g/L - transfusions acceptable

Total bilirubin- less than or equal to 1.5 times the institutional upper limits of normal

Aspartate aminotransferase (AST)serum glutamic oxaloacetic transaminase(SGOT) and alanine aminotransferase (ALT)serum glutamic pyruvic transaminase(SGPT) - less than or equal to 2.5 times the institutional upper limits of normal

Creatinine or Creatinine clearance- less than or equal to 1.5 times the institutional upper limits of normal or greater than or equal to 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

Recovered from any toxicity from surgery or radiotherapy

Must be willing to travel from their home to the National Institutes of Health (NIH) for follow-up visits

Able and willing to follow instructions and conform to protocol.

Patients may have had no other active malignancy within the past 2 years with the exception of non-melanoma skin cancer and superficial bladder carcinoma

No history of myocardial infarction within the past 6 months, uncontrolled congestive heart failure (CHF) or uncontrolled angina pectoris

Patients must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 2 months after completion.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Present clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) brain scan.

Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Persistent systolic blood pressure greater than or equal to 170 mmHg or diastolic blood pressure greater than or equal to 100 mmHg.

Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with docetaxel, bevacizumab, and/or the combination.

Proteinuria, as demonstrated by a urine, protein, creatinine (UPC) ratio greater than or equal to 1.0 at screening, required to be assessed if urine dipstick is greater than or equal to 1+.

Urine protein should be screened by urine analysis for Urine Protein Creatinine (UPC) ratio. For UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment. Note: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using one of the following formula:

* [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL
* [(urine protein) x 0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

Therapeutic anticoagulation with coumadin, heparins, or heparinoids.

Greater than Grade 2 peripheral neuropathy at baseline.

History of transient ischemic attacks (TIA) or cerebrovascular accident (CVA) within the past 2 years.

History of allergic reaction to docetaxel, prednisone, thalidomide and/or bevacizumab or related products.

Patients who are on concurrent investigational agent(s)

Patients who are unable to ingest oral medication.

INCLUSION OF WOMEN AND MINORITIES

Men of all races and ethnic groups are eligible for this trial. Every effort will be made to recruit minorities in this study. Women are ineligible for this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-04-19 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horwitz SB. Taxol (paclitaxel): mechanisms of action. Ann Oncol. 1994;5 Suppl 6:S3-6. PMID 7865431
- [Background] McDonnell TJ, Troncoso P, Brisbay SM, Logothetis C, Chung LW, Hsieh JT, Tu SM, Campbell ML. Expression of the protooncogene bcl-2 in the prostate and its association with emergence of androgen-independent prostate cancer. Cancer Res. 1992 Dec 15;52(24):6940-4. PMID 1458483
- [Background] Berchem GJ, Bosseler M, Sugars LY, Voeller HJ, Zeitlin S, Gelmann EP. Androgens induce resistance to bcl-2-mediated apoptosis in LNCaP prostate cancer cells. Cancer Res. 1995 Feb 15;55(4):735-8. PMID 7850782
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0257.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Main Cohort - Prostate Cancer | Expansion Cohort - Prostate Cancer
Started | 60 | 13
Completed | 57 | 12
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Cohort - Prostate Cancer | Expansion Cohort - Prostate Cancer | Total
Number analyzed (Participants) | 60 | 13 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 8 | 37
  >=65 years | 31 | 5 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.35 (7.81) | 63.31 (8.74) | 64.98 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 13 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 56 | 12 | 68
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 51 | 11 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 13 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Prostate-specific Antigen (PSA) Response
Description: PSA response was assessed by the PSA Consensus Criteria. PSA decline is defined as a decline in PSA of at least 50% with no other evidence of disease progression.
Time Frame: 21.6 months
Population: The main cohort was designed to evaluate clinical progression and the expansion cohort was designed to evaluate immune response. Thus the expansion cohort is not included here.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 60
Participants | 52

2. Primary Outcome: Immune Response
Description: Cellular immune response and cytokines were evaluated after two cycles of therapy in the expansion cohort. Those cycles included treatment with bevacizumab and docetaxel as a pre-medication.
Time Frame: 6 weeks
Population: Cellular immune response and cytokines were not analyzed as the study outcomes were concentrated on the dual-anti-angiogenesis inhibition properties of the regimen and not immunomodulatory changes.
Arm/Group | Expansion Cohort - Prostate Cancer
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort - Prostate Cancer | Expansion Cohort - Prostate Cancer
Number analyzed (Participants) | 60 | 13
Participants | 60 | 13

4. Secondary Outcome: Time to Progression Using Bubley Criteria
Description: Time to disease progression was based on the Prostate-Specific Antigen (PSA) Working Group 1 Criteria (Bubley Criteria) and standard Response Evaluation Criteria in Solid Tumors (RECIST) for measurable disease. Per the criteria, investigators report at a minimum a PSA decline of at least 50% and this must be confirmed by a second PSA value 4 or more weeks later. Patients may not demonstrate clinical or radiographic evidence of disease progression during this time period.
Time Frame: up to 40 months
Population: Per protocol, time to progression using Bubley Criteria was not assessed for the expansion cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 60
Months | 18.3 [0 to 40]

5. Secondary Outcome: Disease Progression by Clinical and Radiographic Criteria Without the Use of Prostate-Specific Antigen (PSA)
Description: Clinical and radiographic response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking s reference the smallest sum LD since the treatment started. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded or the appearance of one or more new lesions.
Time Frame: up to 34 months
Population: Only 33/60 participants had measurable disease and were evaluable for this outcome measure.
  Per protocol, disease progression by clinical and radiographic criteria without the use of PSA was not assessed for the expansion cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 33
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 19
  Stable Disease (SD) | 11
  Progressive Disease (PD) | 1

6. Secondary Outcome: Number of Participants Who Died After a Follow Up of 34 Months Following Treatment
Description: From on study date to date of death at 34 months.
Time Frame: 34 months
Population: Per protocol, this outcome was not assessed for the expansion cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 60
Participants | 38

7. Secondary Outcome: Plasma Concentrations of Docetaxel and Thalidomide and Clinical Activity or Toxicity
Description: The analysis will be performed using a validated method based on liquid chromatography with mass-spectrometric detection.
Time Frame: Pre-dose on C1D1, 5 minutes before the end of infusion, and 15, and 30 minutes, and 1, 2,4,8, and 24 hours after the end of infusion
Population: The outcome was not assessed as the analysis of plasma bevacizumab concentrations was the main pharmacokinetic secondary outcome in the study. The plasma levels of docetaxel and thalidomide (without bevacizumab) had minimal significance in this study. Analysis of plasma concentrations of docetaxel and thalidomide will not be done.
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With a Significant Increase in Circulating Apoptotic Endothelial Cell (CAEC) Level
Description: The assay utilized has no standard curve. Categorizing patients with ≥ 75% PSA decline in one group and < PSA decline in another group, every patient is their own control with comparison of CAEC at baseline vs. 6 weeks (after two cycles of treatment). Blood is drawn from the patient and a million viable mononuclear cells are counted and then it is determined how many CAECs are in the specimen. The cell count is then compared from baseline to post 2 cycles of treatment. Thus, "significant increase" is dependent upon this comparison and varies between patients.
Time Frame: Baseline and at 6 weeks (after two cycles of treatment)
Population: Only 17/60 participants were evaluable for this outcome. Per protocol CAECs were not assessed in the expansion cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Main Cohort - Particpants With ≥75% PSA Decline; Main Cohort - Particpants With <75% PSA Decline: Docetaxel 75 mg/m^2 intravenously over 60 minutes on cycle 1 day 1 repeated every 21 days. Thalidomide 200 mg by mouth daily throughout the cycle. Prednisone 10 mg by mouth daily throughout the cycle. Bevacizumab 15 mg/kg intravenously on cycle 1 day 1 every 21 days.
Arm/Group | Main Cohort - Particpants With ≥75% PSA Decline | Main Cohort - Particpants With <75% PSA Decline
Number analyzed (Participants) | 14 | 3
Participants | 14 | 0
Statistical Analysis 1: Comparison: Main Cohort - Particpants With ≥75% PSA Decline vs Main Cohort - Particpants With <75% PSA Decline; Test type: Superiority or Other; p = .02, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Analyze the Patients Genotype With Regard to Cytochrome P450 2C19 Polymorphism and Correlate That With Pharmacokinetics and Efficacy
Description: Single nucleotide polymorphisms in genes that play an important role in eliminations pathways for docetaxel (in the CYP3A4 and CYP3A5 genes) and thalidomide (CYP2C19) will be evaluated.
Time Frame: Patient entry onto the study
Population: The outcome was not assessed as the clinical significance of cytochrome P450 2C19 polymorphism in angiogenesis is undetermined. This analysis will not be pursued.
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 0

10. Secondary Outcome: Usefulness of Dynamic Magnetic Resonance Imaging (MRI) to Monitor the Progression of Bony and Soft Tissue Disease in Metastatic Prostate Cancer
Description: Target lesions in the bone or soft tissues will be identified from the participant computed tomography (CT) scan. Dynamic MRI will be performed after the intravenous administration of 0.1 mmol/kg of Gadolinium chelate. Progression is defined by the RECIST criteria and is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment starts or the appearance of new lesions.
Time Frame: Baseline and at 3 month intervals until progression
Population: The outcome was not assessed as the functionality of dynamic MRI in prostate cancer was poor at the time of this study. Earlier prostate MRI techniques suffered from poor sensitivity and specificity for monitoring progression.
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 0

11. Secondary Outcome: Changes in the Molecular Markers of Angiogenesis (Including, But Not Limited to Serum and Urine Vascular Endothelial Growth Factor (VEGF)) Before and After Administration of Docetaxel, Prednisone, Thalidomide and Bevacizumab
Time Frame: Baseline and monthly
Population: The outcome was not assessed. In the study, assessment of circulating apoptotic endothelial cells was the main outcome evaluated for assessing the treatment's antiangiogenic activity. Changes in the molecular markers of angiogenesis will not be pursued.
Arm/Group | Main Cohort - Prostate Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 37 months
Arm/Group | Main Cohort - Prostate Cancer | Expansion Cohort - Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 35/60 | 1/13
Serious Adverse Events (participants affected / at risk) | 48/60 | 4/13
Other Adverse Events (participants affected / at risk) | 60/60 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort - Prostate Cancer (N=60) | Expansion Cohort - Prostate Cancer (N=13)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 2 (3) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac arrhythmia - Other, Specify, new onset of A. fib (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac general - Other, Specify, aortic dissection (Cardiac disorders) | 1 (1) | 0 (0)
Death not associated with CTCAE term::Death NOS (General disorders) | 9 (9) | 0 (0)
Death not associated with CTCAE term: Death Progression NOS (General disorders) | 25 (25) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L), fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hemoglobin (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hemorrhage, GI: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Upper GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) : urinary tract NOS
Infection with normal ANC or Grade 1 or 2 neutrophils:Abdomen NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Anal/perianal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 4 (4) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC: Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neurology-Other (somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AG) (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Cardiac/heart (Cardiac disorders) | 1 (1) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Proteinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Supraventricular and nodal arrhythmia::Nodal/Junctional (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 0 (0)
Vessel injury-artery: Aorta (Vascular disorders) | 1 (1) | 0 (0)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0) — with grade 3 or 4 neutrophils) (ANC <1.0X10e9/L)Skin:cellulitis
Infection (documented clinically or microbiologically) with Grade 3 or 4 (Infections and infestations) | 0 (0) | 1 (1) — neutrophils (ANC1.0x10e9/L) : urinary tract NOS
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection with unknown ANC: Wound (Infections and infestations) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (acute kidney injury; chronic kidney disease) (Renal and urinary disorders) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Infection - Other (sepsis) (Infections and infestations) | 1 (1) | 0 (0)
Death not associated with CTCAE term: Death, Progression NOS (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort - Prostate Cancer (N=60) | Expansion Cohort - Prostate Cancer (N=13)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 14 (20) | 2 (8)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 14 (28) | 2 (6)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 41 (97) | 5 (7)
Alkaline phosphatase (Metabolism and nutrition disorders) | 12 (19) | 2 (8)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (4) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 7 (7) | 2 (2)
Anorexia (Gastrointestinal disorders) | 7 (8) | 3 (4)
Ataxia (incoordination) (Nervous system disorders) | 6 (10) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (6) | 1 (4)
Bladder spasms (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood/Bone marrow - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Anemia; neutropenia
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 7 (9) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 22 (36) | 3 (4)
Cardiac arrhythmia - Other, Specify, (Cardiac disorders) | 3 (3) | 1 (1) — bradycardia; cardiac; tachycardia; vasovagal episode
Cardiac general - Other, Specify, (Cardiac disorders) | 3 (3) | 2 (2) — chest discomfort or no CP; diastolic murmur; tachycardia; chest tightness
Chelitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coagulation - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Bleeding at injection site
Cognitive disturbance (Nervous system disorders) | 3 (3) | 1 (1)
Constitutional Symptoms-Other (Specify,_____) (General disorders) | 3 (4) | 0 (0) — night sweats; weight loss
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 3 (3) | 0 (0)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (7) | 1 (1)
Dental: periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental: teeth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dermal change lymphedema, phlebolymphedema (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 21 (24) | 6 (9)
Dizziness (Nervous system disorders) | 17 (22) | 3 (3)
Dry eye syndrome (Eye disorders) | 6 (7) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 22 (22) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 26 (37) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 13 (17) | 5 (6)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 52 (76) | 11 (23)
Febrile Neutropenia (Infections and infestations) | 13 (15) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC < 1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (General disorders) | 6 (9) | 2 (2) — (in the absence of neutropenia, where neutropenia is defined as AGC<1.0x10e9/L)
Flu-like symptoms (Immune system disorders) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 3 (3) | 5 (7) — anorexia; early satiety; GI-disturbance-related to dairy; gingivitis-infection; L abdominal mass; melena; mucositis; stomach cramps secondary to constipation; abdominal bloating; teeth changes color
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (8) | 1 (5)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 31 (33) | 5 (5)
Hearing: patients with/without baseline auidgram and not enrolled in a monitoring program) (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hemoglobinuria (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemolysis (e.g., immune hemolytic anemia, drug related hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, GI: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 5 (5) | 0 (0)
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage, GU: Urethra (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 19 (32) | 5 (7)
Hemorrhage, pulmonary/upper respiratory: Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 6 (7) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 17 (20) | 4 (5)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 7 (7) | 1 (1)
Incontinence, anal (Gastrointestinal disorders) | 5 (5) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0x10e9/L): Abdomen NOS
Infection - Other, Specify (Infections and infestations) | 3 (4) | 2 (3) — bronchitis; left great toe infection; left eye conjunctiva; paronychia R great toe; URI-cough & wheezing; URI-sore throat; upper respiratory infection
Infection with normal ANC or Grade 1 or 2 neutrophils: Anal/perianal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils: Conjuctiva (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Larynx (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Middle ear (otitis media) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Muscle (infection myositis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Nerve-peripheral (Infections and infestations) | 1 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Nose (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:paranasal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Sinus (Infections and infestations) | 5 (5) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils:Ungual (nails) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:Upper airway NOS (Infections and infestations) | 2 (2) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils:Urinary tract NOS (Infections and infestations) | 3 (3) | 0 (0)
Infection with unknown ANC::Middle ear (otitis media) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC:Sinus (Infections and infestations) | 2 (2) | 1 (1)
Infection with unknown ANC::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Soft tissue NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Ungual (nails) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1) | 2 (2)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 2 (2) | 2 (2)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 36 (74) | 11 (27)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Keratitis (corneal inflammatory/corneal ulceration) (Eye disorders) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lymphatics - Other (Specify) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — small upper lobe nodes
Lymphopenia (Blood and lymphatic system disorders) | 37 (160) | 9 (35)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 7 (8) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 0 (0)
Metabolic/Laboratory - Other (Specify) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — LDH, high
Mood alteration-agitation (Nervous system disorders) | 2 (2) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1) | 2 (2)
Mood alteration::Depression (Nervous system disorders) | 6 (9) | 1 (2)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 6 (7) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Espophagus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 3 (4) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Muscle weakness, generalized or specific area (not due to neuropathy)::Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::trunk (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0)
Musculoskeletal/Soft tissue - Other (Specify,) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 29 (31) | 7 (9)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (10) | 4 (9)
Neurology-Other (Specify,______) (Nervous system disorders) | 10 (14) | 0 (0)
Neuropathy - cranial::CN IX Motor-pharynx; sensory-ear, pharynx tongue (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy - cranial::CN V Motor-jaw muscles; sensory-facial (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy - cranial::CN VIII Hearing and balance (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 9 (11) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 45 (65) | 6 (9)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 35 (71) | 11 (29)
Ocular/Visual-Other (Specify,___) (Eye disorders) | 3 (3) | 2 (3) — conjunctival injection; decreased visual acuity; diplopia; eye tearing; mucus discharge for eyes; near vision problem
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 (0) | 1 (1)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 2 (2) | 0 (0)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 12 (24) | 1 (3)
Pain-Other (Specify,R leg pain; shoulder pain; tooth pain; jaw) (General disorders) | 13 (18) | 2 (2) — (R) hip/leg pain; finger tips; heel pain; jaw w/hx of ONJ; L calf; L lower jaw sensitivity; left knee; left shoulder pain; lower back pain; pain-(L) elbow and groin; pain-(L) shoulder; R ear pain; R arm pain-mid arm (known bone mets); R hip pain
Pain: Abdomen NOS (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pain: Back (Musculoskeletal and connective tissue disorders) | 11 (12) | 6 (6)
Pain::Cardiac/heart (Cardiac disorders) | 1 (2) | 0 (0)
Pain::Chest wall (Cardiac disorders) | 2 (2) | 1 (1)
Pain::Chest/thorax NOS (Cardiac disorders) | 2 (2) | 0 (0)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Pain: Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 7 (9) | 3 (5)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1)
Pain::Oral cavity (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pain::Oral gums (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Pain NOS (General disorders) | 1 (1) | 0 (0)
Pain::Pelvis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain::Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Perforation, GI::Colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2) | 1 (1)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 24 (54) | 5 (19)
Platelets (Blood and lymphatic system disorders) | 13 (21) | 2 (5)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 15 (20) | 4 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 10 (17) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, ) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13 (14) | 7 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11 (14) | 0 (0)
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 3 (3) | 0 (0) — hematuria; nephrotic syndrome
Salivary gland changes/saliva (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scleral necrosis/meli (Eye disorders) | 1 (1) | 0 (0)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 (14) | 2 (5)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 8 (15) | 1 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 33 (38) | 8 (9)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (4) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 8 (8) | 0 (0)
Ulcer, GI: Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 7 (7) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (3) | 0 (0)
Vasovagal episode (Cardiac disorders) | 2 (2) | 0 (0)
Vessel injury-vein: Extremity-lower (Vascular disorders) | 1 (1) | 0 (0)
Vessel injury-vein: Other NOS (Vascular disorders) | 1 (1) | 1 (1)
Vision-blurred vision (Eye disorders) | 9 (10) | 0 (0)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (4)
Watery eye (epiphora, tearing) (Eye disorders) | 26 (32) | 7 (8)
Weight gain (General disorders) | 3 (3) | 2 (3)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Weight loss (General disorders) | 10 (15) | 1 (2)
Dermatology/Skin-Other (Specify,_____) (Skin and subcutaneous tissue disorders) | 9 (14) | 0 (0) — cellulitis; ecchymosis; lip-abscess; oral leukopenia; RLE sunburn; rash; decubitus ulcer R buttock; ecchymosis at injection sites; fingers blister; folliculitis; generalized erythema; peeling in sole
Hemoglobin (Metabolism and nutrition disorders) | 35 (153) | 8 (23)
Hemorrhage/Bleeding - other (Specify) (Blood and lymphatic system disorders) | 6 (8) | 0 (0) — conjunctiva hemorrhage/right eye; ecchymosis; epistaxis; hematochezia; intermittent hard stool with blood-hematochezia; bleeding to Lovenox sites; bleeding to lower lip
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 46 (64) | 8 (10)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically): dental tooth (Infections and infestations) | 1 (1) | 0 (0) — with grade 3 or 4 neutrophils (ANC,1.0x10e9/L)
Infection (documented clinically or microbiologically): upper airway NOS (Infections and infestations) | 2 (2) | 0 (0) — with grade 3 or 4 neutrophils (ANC<1.0x10e9/L)
Infection (documented clinically or microbiologically): urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0) — with grade 3 or 4 neutrophils (ANC<1.0x10e9/L)
Infection (documented clinically or microbiologically): cellulitis (Infections and infestations) | 1 (1) | 0 (0) — with grade 3 or 4 neutrophils (ANC<1.0x10e9/L)
Obstruction, GU: Ureter (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstruction, GU: Urethra (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT00089609/Prot_SAP_ICF_000.pdf